CLINICAL TRIAL: NCT05124041
Title: Thromboelastometry Guided Transfusion Protocol Versus Standard Care in Acute-on-Chronic Liver Failure with Bleeding: a Prospective Intervention Trial
Brief Title: Goal-Directed Hemostatic Resuscitation Trial in ACLF Induced Coagulopathy
Acronym: GOODHEART-ACLF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PGI/IEC/2020/000268; PGI/IEC/2024/EIC000462 27.3.24 (Other: PGIMER Institutional review board)
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Acute on Chronic Liver Failure; Variceal Hemorrhage; Cirrhosis, Liver; Thromboelastometry; Thrombosis;Portal
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: 260 patients having ACLF with bleeding will be randomized into two groups. One will be treated conventionally, i.e. using clinical judgement and conventional coagulation tests, the other treated using a ROTEM-based algorithm
  Revised Eligibility criteria as per Baveno VII ACLF with variceal bleeding with any indication for blood component transfusion as below
  Indications for transfusion in either arm are
  1. Multiple sites of bleed e.g. diffuse mucosal ooze, post EVL ulcers, diffuse portal hypertensive gastropathy, etc which are associated with coagulation dysfunction against a background of portal hypertensive bleeding
  2. Failure to control bleeding
  3. Early rebleeding
  4. Active bleeding on endoscopy with refractory variceal bleeding, need for balloon tamponade or self expandable metal stents (SEMS)
  5. At the time of bridge therapy to a more definite treatment such as PTFE covered TIPS.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ROTEM-arm (Experimental): Treatment of significant blood loss using point-of-care testing of whole blood viscoelasticity (ROTEM) monitoring coagulopathy or hyperfibrinolysis
  Interventions: Diagnostic Test: Rotational thromboelastometry
- Control-arm (Active Comparator): Treatment of significant blood loss conventionally, ie. using clinical judgement and conventional coagulation tests, such as prothrombin time (as international normalized ratio, INR), activated partial thrombin time (APTT), fibrinogen in plasma
  Interventions: Diagnostic Test: Rotational thromboelastometry

INTERVENTIONS:
Diagnostic Test: Rotational thromboelastometry — ROTEM-guided protocol of hemostatic resuscitation

SUMMARY:
In this project, we plan to evaluate whether a new, rotational thromboelastometry-guided algorithm (ROTEM) to guide hemostatic resuscitation decreases the use of allogeneic blood products, the total amount of bleeding, transfusion related side effects, thromboembolic complications and costs. Its effect on each patient's post-operative hemostatic profile is also measured.

We plan to enroll 260 patients having ACLF with variceal bleeding randomized into two groups: one will be treated conventionally using clinical judgement and standard coagulation tests such as prothrombin time, platelet count, etc. the other treated using a ROTEM-based algorithm. They will be followed for development of rebleeding, complications of transfusion and any signs of infection after hospitalization

There will be a 'no intervention' group with well controlled bleeding who will undergo VETs but not be offered coagulation correction prophylactically in accordance with the Baveno VII consensus. This control group will be followed up in parallel with the main intervention groups.

The ROTEM or SCT based correction will only be offered to patients who have high risk for rebleeding/ failure to control bleeding/ active bleeding at endoscopy/ need SEMS/TIPS and such individuals will be randomized to 2 arms ROTEM vs SCT, with 130 in each arm.

DETAILED DESCRIPTION:
Patients with acute-on-chronic liver failure (ACLF) have coagulation failure in the setting of systemic inflammatory syndrome (SIRS), sepsis and extra-hepatic organ failures. The utility of thromboelastography/thromboelastometry currently has unvalidated clinical benefit in the assessment and reversal of coagulopathy among cirrhotic patients as compared to standard coagulation testing.Need for periprocedural blood transfusion is still high in patients with decompensated cirrhosis or ACLF who present with major bleeding. Allogeneic blood transfusion may be detrimental in patients with cirrhosis, due to volume overload and acute lung injury. Viscoelastic testing of global coagulation such as thromboelastometry has been proposed as a superior tool to rapidly diagnose and help guide resuscitation with blood products. In prior studies, we have clarified the pathophysiology of hemostasis in relation to the evidence of sepsis in liver disease and described the accuracy of various available laboratory tests in assessment of these patients. We have described the role of endogenous heparinoids in severe alcoholic hepatitis and the pathogenesis of the coagulation defect in ACLF. We determined the influence of sepsis on coagulation disorders in ACLF patients, to correctly identify the type and optimal quantity of blood product requirement in at risk patients.

ELIGIBILITY:
Patient with ACLF with variceal bleeding is eligible for the study if one or more of the criteria are met following primary endoscopic intervention.

1. Multiple sites of bleed e.g. diffuse mucosal ooze, post EVL ulcers, diffuse portal hypertensive gastropathy, etc which are associated with coagulation dysfunction against a background of portal hypertensive bleeding
2. Failure to control bleeding
3. Early rebleeding
4. Active bleeding on endoscopy with refractory variceal bleeding, need for balloon tamponade or self expandable metal stents (SEMS)
5. At the time of bridge therapy to a more definite treatment such as PTFE covered TIPS.

If one of the above criteria is met, then the patient is enrolled provided they meet the criteria below.

Inclusion Criteria:

* Age 18-65 years
* ACLF, as diagnosed by CANONIC/ APASL criteria .
* Upper gastrointestinal bleeding

Exclusion Criteria:

* Current therapy: Recent blood or blood component transfusion in the last 2 weeks.
* HIV positive/ AIDS patients
* Patients requiring antiplatelet therapy,
* Renal insufficiency requiring dialysis
* Active malignancy within the last 5 years
* Patient with other neurological disease and metabolic disorders, unbalanced heart failure and/or respiratory failure or end-stage renal disease
* Administration of anticoagulants, antifibrinolytics,
* Not willing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with clinical control of bleeding | 24 hours
  Clinical control of bleeding at 24 hours, at Day 5 and day 42
Number of participants with clinical control of bleeding | 5 days
  Clinical control of bleeding at 24 hours, at Day 5 and day 42
Number of participants with clinical control of bleeding | 42 days
  Clinical control of bleeding at 24 hours, at Day 5 and day 42

SECONDARY OUTCOMES:
Duration of Intensive care admission | 30 days after bleeding episode treated by transfusion protocol
Duration of hospital stay | 30 days after bleeding episode treated by transfusion protocol
Number of Participants with Transfusion-related side effects | 30 days after bleeding episode treated by transfusion protocol
Number of Participants with Thromboembolic events | 30 days after bleeding episode treated by transfusion protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Choose Any State/Province, India

IPD SHARING:
Plan to Share IPD: Undecided